CLINICAL TRIAL: NCT07274306
Title: Incidence, Treatment of and Outcome of Acute Mesenteric Ischemia in the Region of Västra Götaland, 2000-2023 - a Retrospective Observational Study
Brief Title: Incidence, Treatment and Outcome After Acute Mesenteric Ischemia in the Region of Västra Götaland, 2000-2023.
Acronym: AMIGO
Status: Active, not recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Gothia Forum - Center for Clinical Trial (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Hanna de la Croix, MD, PhD, Sahlgrenska University Hospital
Other Study IDs: 2024-04585-01
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Mesenteric Artery Ischemia
Keywords: Acute mesenteric ischemia; Mesenteric ischemia; Intestinal ischemia; Population-based cohort; Epidemiology; Incidence; Mortality; Mesenteric arterial occlusion; Sweden / Västra Götaland
MeSH Terms: conditions — Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VG Region patients with AMI diagnosis 2000-2023: A cohort of all patients who were discharged with the diagnosis acute mesenteric ischemia (ICD-10: K55.0 or K55.9) in the Västra Götaland region of Sweden between 2000-01-01 and 2023-12-31.

SUMMARY:
The goal of this retrospective observational study is to describe the incidence and outcome of patients diagnosed with acute mesenteric ischemia (AMI) in the Västra Götaland region of Sweden between 2000-2023. The main questions it aims to answer are:

* What was the observed incidence and outcome, and how did it change during the time period?
* How did socioeconomic factors influence incidence and outcome of AMI?
* What main surgical approaches were selected for these patients?
* What was the distribution of anticoagulant use in the cohort, and what effect did the introduction of new oral anticoagulants (NOAC) have on incidence and mortality in AMI?
* What was the prevalence of Short Bowel Syndrome (SBS) after surgical intervention?

Participants were obtained from the regional diagnosis registry. Additional datapoints were obtained from the Swedish statistics bureau and pharmaceutical registers.

ELIGIBILITY:
Inclusion Criteria:

* all patients discharged from hospital with acute mesenteric ischemia (ICD K55.0 and K55.9)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inhabitants of the Västra Götaland region in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 2446 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute mesenteric ischemia | Year 2000-2023
  Annual incidence rate of acute mesenteric ischemia per 100,000 person-years in the Västra Götaland region.
Mortality from acute mesenteric ischemia | 30 days, 90 days, 1 year.
  All-cause mortality within up to 1 year of AMI diagnosis.

SECONDARY OUTCOMES:
Temporal trends in incidence and mortality | Year 2000-2023
  Change over time in incidence and mortality, including before and after introduction of non-vitamin K antagonist oral anticoagulants (NOACs).
Socioeconomic determinants of incidence and outcome | Year 2000-2023
  Association between SES indicators (income, education, immigration status, geographic distance to care) and risk of AMI or mortality.
Surgical management strategy | Year 2000-2023
  Proportion of patients undergoing bowel resection, revascularization (open or endovascular), or non-operative management.
Prevalence of Short Bowel Syndrome (SBS) | Within 1 year of surgical intervention
  Number and percentage of patients developing SBS (ICD-10 K91.2 and K90.8) after AMI.
Anticoagulant use patterns | At AMI diagnosis; trends from 2000-2023
  Proportion of patients using vitamin-K antagonists, NOACs, antiplatelet therapy, or no anticoagulation; association with incidence and survival.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Sahlgrenska hospital/Östra hospital, Gothenburg, Västra Götaland County
  - Sahlgrenska University Hospital, Gothenburg

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Due to Swedish data protection legislation and ethical restrictions, the de-identified dataset cannot be made publicly available. Only aggregated results will be published.